CLINICAL TRIAL: NCT03088722
Title: Task-sharing to Expand Access to Contraceptive Implants: A Study Comparing Implant Provision by Community Health Extension Workers With Nurses and Midwives in Nigeria
Brief Title: A Study Comparing Implant Provision by Community Health Extension Workers With Nurses and Midwives in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Stopes International (Other)
Collaborators: Population Council (Other); GRM Futures Group (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E2331
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Contraception
Keywords: Contraceptive implant; Task sharing; Nigeria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community health extension workers (Experimental): Community health extension workers providing contraceptive implants
  Interventions: Other: Training CHEWs to provide contraceptive implants
- Nurses and midwives (No Intervention): Nurses and midwives providing contraceptive implants (existing care)

INTERVENTIONS:
Other: Training CHEWs to provide contraceptive implants — Training CHEWs to provide contraceptive implants
  Arms: Community health extension workers

SUMMARY:
This proposed study, to be run by Marie Stopes International Organisation Nigeria (MSION) will investigate whether Community Health Extension Workers (CHEWs) in Nigeria can insert and remove contraceptive implants to the same level of safety and quality as a nurse or midwife, and whether this is acceptable to their clients and colleagues. The study will also document feasibility issues which would be relevant to any future national programmatic scale-up.

ELIGIBILITY:
Inclusion Criteria:

* facilities are located with 20km of a referral facility
* facilities - facility staff are willing to participate, e.g. willingness to conduct family planning awareness-raising activities, willing to maintain project records
* facilities - selected provider at each facility expects to be in the facility for the 12-month period of client recruitment
* clients - women present to attending facilities and request a contraceptive implant

Exclusion Criteria:

* facilities - involved in overlapping interventions

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7903 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | Day of implant insertion
  Any adverse event recorded by the health provider or the client on the day of the procedure

SECONDARY OUTCOMES:
Quality of implant provision | Day of implant insertion
  Supervisor-recorded quality of service provision, which includes includes both clinical dimensions, such as cleanliness, and non-clinical dimensions, such as taking a client focused approach and being responsive to client needs
Acceptability of service provision | Day of implant insertion
  Client-reported views of implant provision
Adverse events | Up to 14 days post insertion
  Any adverse event recorded by the health provider at the time of implant insertion or reported by the client on the day of the procedure or up to 14 days after the procedure

REFERENCES:
- [Derived] Reiss K, Penfold S, Alabi O, Ali M, Hopkins K, Ngo TD, Odogwu K, Douthwaite M, Ezire O, Udoh U, Effiom E, Munroe ES. Safety, Quality, and Acceptability of Contraceptive Subdermal Implant Provision by Community Health Extension Workers Versus Nurses and Midwives in Nigeria: Protocol for a Quasi-Experimental, Noninferiority Study. JMIR Res Protoc. 2018 Mar 2;7(3):e67. doi: 10.2196/resprot.8721. PMID 29500162